CLINICAL TRIAL: NCT07096999
Title: SPECT/CT Imaging for Dosimetry in 177Lu-PSMA-617 (Pluvicto) Therapy
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UMCC 2024.070; NCI-2025-01555 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00257753 (Other: University of Michigan Comprehensive Cancer Center); R01CA289631 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration-Resistant Prostate Carcinoma
Keywords: Prostate Cancer; 177Lu; PSMA; mCRPC; Radioligand Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational: Patients receive standard care Pluvicto and undergo Lu-177 SPECT/CT scans on study. Patients may also undergo optional 99mTc-SC SPECT/CT scan for bone marrow dosimetry prior to cycle 1. In addition, patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being performed to establish the association between absorbed dose to tumor and response and absorbed dose to normal organs and toxicity following Lu177-PSMA radioligand therapy

ELIGIBILITY:
Inclusion Criteria:

* * 177Lu-617 PSMA treatment scheduled for mCRPC

  * Clinically stable as determined by the nuclear medicine clinicians
  * Male
  * ≥ 18 years of age
  * Willing and able to provide informed consent

Exclusion Criteria:

* Patients who are unable to lie flat on the imaging systems long enough to permit imaging protocols to be performed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mCRPC undergoing 177Lu-PSMA-617 treatment at the University of Michigan
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2031-01-23 (Estimated); Study Completion 2031-01-23 (Estimated)

PRIMARY OUTCOMES:
Response and toxicity following 177Lu-RLT | Up to 4 years
  Association between absorbed dose and effect (response/toxicity) following 177Lu-RLT

SECONDARY OUTCOMES:
Build and test models | Up to 4 years
  Build and test models for predicting therapy delivered absorbed dose from pre-therapy PET imaging/non-imaging biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Yuni K Dewaraja, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided